CLINICAL TRIAL: NCT01513187
Title: Phase I/II Prospective, Open Label and Multicentric Clinical Trial to Determine the Recommended Dose (Phase I) and Efficacy of Pazopanib in Combination With Interferon Alfa 2-A (Phase II), in Patients With Advanced Renal Cell Carcinoma
Brief Title: Pazopanib in Combination With Interferon Alfa 2-A, in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2010-01
Record Dates: First submitted 2012-01-10; First posted 2012-01-20 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2020-03

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: Advanced renal cell carcinoma; SOGUG; Pazopanib; Pazopanib in combination with interferon alpha 2A
MeSH Terms: interventions — pazopanib; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib + interferon (Experimental): Five levels of pazopanib in different doses: 400, 600 and 800 mg / day and interferon alfa 2-A 3, 6 and 9 MIU three times a week, in cycles of 28 days.
  Treatment will continue until disease progression, unacceptable toxicity, non-compliance or withdrawal of consent by the patient
  Interventions: Drug: Pazopanib + interferon alpha 2A

INTERVENTIONS:
Drug: Pazopanib + interferon alpha 2A — Five levels of pazopanib in different doses: 400, 600 and 800 mg / day and interferon alfa 2-A 3, 6 and 9 MIU three times a week, in cycles of 28 days.
  Treatment will continue until disease progression, unacceptable toxicity, non-compliance or withdrawal of consent by the patient

SUMMARY:
Phase I / II, open, prospective, multicenter single-arm, Clinical Trial in two stages: in the first stage it will determine the optimal dose of the combination of pazopanib and interferon alfa-A2 in the treatment of patients with advanced renal carcinoma and a second stage that will determine the efficacy of this combination measured in terms of response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years.
3. Patients diagnosed histologically clear cell carcinoma of the kidney metastatic or unresectable locally advanced, previously untreated. However, in Phase I may include patients with primary tumors other than renal cell can benefit from these drugs and patients with renal cell carcinoma treated before.
4. Performance status (ECOG) 0-1.
5. Patients must have measurable disease by RECIST criteria V 1.1. Progression should be documented in the two months prior to study entry.
6. Patients may not have received prior treatment with anti-VEGF agents, mTOR inhibitors or cytokines. However, in Phase I may include patients who have received any previous treatment.
7. Paraffin tumor sample should be available and collection of serum from all subjects for biomarker analysis previously and / or during treatment with study medication.
8. Adequate Hematologic, liver and kidney functions.
9. Women of childbearing potential must be using an effective method of birth control (abstinence, any intrauterine device [IUD] published data showing that the expected minimum rate of failure is less than 1% per year, or any other method the published data show that the expected minimum rate of failure is less than 1% per year) before inclusion in the study and continue using it during the same six months after completion. Women of childbearing age should get a negative pregnancy test in urine or serum (minimum sensitivity 25 IU / L or equivalent units of beta fraction of human chorionic gonadotropin [β-HCG]) during the seven days prior to the randomization.
10. Able to swallow oral compound.
11. Willingness and ability to attend scheduled visits, to follow the treatment schedule and to undergo clinical trials and other study procedures

Exclusion Criteria:

1. History of prior malignancies diagnosed or treated over the past 5 years except basal cell skin cancer or prostate cancer incidentally detected previously treated. However, patients with a history of malignancy but free of the disease over the past 5 years, or patients with a history of nonmelanoma skin carcinoma-completely-resected or carcinoma in situ treated successfully can participate in the study .

   In Phase I, patients diagnosed with other previous or concomitant malignant diseases can be included.
2. Presence of metastases in the central nervous system (CNS) or leptomeningeal carcinomatosis, except for patients with previously treated CNS metastases, asymptomatic and have not needed corticosteroids or anticonvulsant drugs in the 3 months prior to administering the first dose of the drug under study. Only is required CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) if clinically indicated or if the individual has a history of CNS metastases.
3. Clinically significant gastrointestinal disorders may increase the risk of gastrointestinal bleeding including, but not limited to:

   Active peptic ulcer disease Known metastatic lesions with probable intraluminal bleeding Inflammatory bowel disease (ulcerative colitis, Crohn's disease) or other gastrointestinal disorders with increased risk of perforation History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days before the start of study treatment.
4. Clinically significant gastrointestinal abnormalities may affect the absorption of the investigational product such as but not limited to:

   Malabsorption syndrome Major resection of the stomach or small intestine Grade 3 diarrhea
5. Patients with active infection or other disease or serious medical condition.
6. Prolongation of the corrected QT wave (QTc)> 480 ms on baseline ECG according to the Bazett formula.
7. Subjects with a history of one or more of the following cardiovascular disease in the last 6 months prior to the inclusion in the study:

   Angioplasty or stent placement Myocardial infarction Unstable Angina Coronary bypass surgery Symptomatic peripheral vascular disease Congestive heart failure Class II, III or IV New York Heart Association (NYHA)
8. Poorly controlled hypertension [defined as systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure stress (DBP) ≥ 90 mmHg] while the patient is on antihypertensive therapy.

   Note: the commencement or adjustment of antihypertensive medication it is possible before the patient study start. In the baseline period measure blood pressure at least twice with a minimum interval of 24 hours. The mean values of SBP / DBP in each blood pressure reading should be <140/90 mmHg to include the subject in the study.
9. Background, in the last six months prior to the inclusion of stroke (including transient ischemic attacks), pulmonary embolism or deep vein thrombosis (DVT) untreated.

   Note: may be included subjects with recent DVT who received anticoagulants for at least 6 months.
10. Surgery or trauma in the last 28 days, or minor surgery (eg., Removal of central venous catheter) in the last 7 days prior to inclusion or unhealed wound, fracture, or ulcer.
11. Evidence of active bleeding or bleeding diathesis.
12. Hemoptysis within 6 weeks prior to inclusion.
13. Pregnant or breastfeeding.
14. Any medical condition (eg. Uncontrolled infection), psychiatric or other to be serious and / or unstable and may interfere with the safety of the patient, obtaining informed consent or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) - Phase I | Up to September 2012
  The MTD is defined as the dose at wich two of the patients have experienced dose-limiting toxicity.
Efficacy, response rate (Phase II) | Up to July 2013
  Response rate is defined as the percentage of patients with complete response or partial response confirmed according RECIST v.1.1

SECONDARY OUTCOMES:
Progression free survival | Up to July 2013
  Period between the start of treatment until the day in in wich the progression is confirmed by RECIST guidelines (version 1.1) or death from any cause.
Overall Survival | Up to December 2013
  Period between the start of treatment and date of death from any cause.
Frequency of adverse events | Up to July 2013
  Toxicity evaluation of the combination using the NCI-CTC Criteria version 3.0
Translational Substudy | Up to December 2013
  To analyze the different biomarkers and their variations with clinical outcomes of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier García del Muro, MD, Principal Investigator — Instituto Catalán de Oncología, Hospitalet del Llobregat
Locations (13):
- Spain (13):
  - Instituto Catalán de Oncología, Hospitalet del Llobregat, L'Hospitalet de Llobregat, Barcelona
  - Centro Integral Oncológico Clara Campal, PAU de Sanchinarro, Sanchinarro - Madrid
  - Hospital del Mar, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma
  - Clinica Univ. Navarra, Pamplona
  - Hospital Virgen de la Macarena, Seville
  - Hospital Virgen del Rocio, Seville
  - Hospital Virgen de la Salud, Toledo
  - IVO, Valencia